CLINICAL TRIAL: NCT06002620
Title: Effect of Cricket Enriched Porridge and Nutrition Education on Stunting, Gut Health and Breastmilk Intake of Infants and Young Children in Western Kenya
Brief Title: Healthynsect Child Growth and Health Intervention Study
Acronym: HEALTHYNSECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Masinde Muliro University of Science and Technology (Unknown); Jomo Kenyatta University of Agriculture and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WP2 HEALTHYNSECT
Record Dates: First submitted 2023-07-10; First posted 2023-08-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2023-08

CONDITIONS: Nutrition Status
Keywords: cricket; insect; complementary feeding; gut health; breastmilk intake; 13C sucrose breath test; deuterium oxide; stable isotopes
MeSH Terms: interventions — Standard of Care; Nutrition Assessment; Educational Status

STUDY DESIGN:
Intervention Model Description: The study has four arms namely: Control arm (CA), Enriched nutrition arm (ENA), Nutrition education arm (NEdA) and a Combined Nutrition Education and enriched nutrition (CEdNA).
  Cricket Enriched flour(CEF) - with cricket, maize, millet, mineral and vitamin premix Corn-Soy Blend plus(CSB+) - with mineral and vitamin premix Nutrition Education- with video, face to face session and SMS reminder
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Stratified by sex, randomization was done by a team not participating in the study implementation and the randomization scheme sent directly to the assigned distribution staff The products under investigation are packed in similar containers differentiated by a code number only known to the distribution staff who is equally blinded of the products contents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control arm (CA) (Experimental): A positive control group using an existing nutritional intervention with the known effect will be adopted, so as to meet ethical practice and be able to determine the effect of our new intervention response on the experimental group. The study will use double blinded approach with the control group receiving standard known flour of the supercereal CSB+ adjusted for ages as follows:6-8 months infants receiving 31g daily,9-11 months receiving 47g and 12-24 months receiving 86g to supply 200,300 and 550KCal daily respectively, with both the caregiver and person administering the food will be blinded from the content of the flour.
  Interventions: Dietary Supplement: CSB+
- Enriched nutrition arm (ENA) (Experimental): The study will use a Cricket Enriched flour(CEF) - with 20% cricket (, maize, millet, mineral and vitamin premix with amounts served adjusted to ages as:6-8 months infants receiving 29g daily,9-11 months receiving 44g and 12-24 months receiving 80g to supply 200,300 and 550KCal daily respectively, with both the caregiver and person administering the food will be blinded from the content of the flour.
  Interventions: Dietary Supplement: Enriched nutrition food (CEF)
- Nutrition education arm (NEdA) (Experimental): Combines the control and nutrition education where nutrition education comprises of a video, face to face session and SMS reminder in predetermined regular sessions
  Interventions: Dietary Supplement: CSB+; Behavioral: Nutrition education
- Combined Nutrition Education and enriched nutrition (CEdNA) (Experimental): Combines the Cricket Enriched flour(CEF) and Nutrition education
  Interventions: Dietary Supplement: Enriched nutrition food (CEF); Combination Product: Combined nutrition and education

INTERVENTIONS:
Dietary Supplement: CSB+ — standard care
  Other Names: Standard care
  Arms: Control arm (CA); Nutrition education arm (NEdA)
Dietary Supplement: Enriched nutrition food (CEF) — enriched cricket flour at 20%
  Arms: Combined Nutrition Education and enriched nutrition (CEdNA); Enriched nutrition arm (ENA)
Behavioral: Nutrition education — regular videos, sms reminders and face to face interaction
  Arms: Nutrition education arm (NEdA)
Combination Product: Combined nutrition and education — combined enriched cricket flour and nutrition education
  Arms: Combined Nutrition Education and enriched nutrition (CEdNA)

SUMMARY:
Malnutrition in all its forms is still a problem in resource limited settings including Kenya driven by low diet quality, food preparation and feeding practices including hygiene. Edible insects are currently of interest in alleviating malnutrition due to their energy density, high protein, vitamins and micronutrients (iron, zinc). Among the insects of preference are the crickets which have been shown to encourage the growth of probiotics (Bifidobacterium animalis) which support gut health increasing nutrient absorption and reduces systemic inflammation. Despite the nutritional value of insects and the contribution of cricket to improved gut health, there is limited evidence on the benefit of cricket based complementary food in the reduction of stunting amongst infants and young children. This study aim to determine the effect of integrating two nutrition interventions (cricket enriched porridge with nutrition education) on the infant and young child growth (stunting) and gut health in Alego Usonga Sub-County in Siaya County of rural western part of Kenya.

DETAILED DESCRIPTION:
Malnutrition in all its forms is still prevalent in resource limited settings driven by low diet quality, food preparation and feeding practices including hygiene. Untreated early childhood malnutrition deprives the child from living to full potential, by increasing susceptibility to childhood infections and is life threatening. Insects are currently of interest in alleviating malnutrition due to their energy density, high protein, vitamins and micronutrients (iron, zinc). Crickets positively support growth of probiotics (Bifidobacterium animalis) which support gut health increasing nutrient absorption and reduces systemic inflammation. Single nutrition interventions are confirmed to be less effective in reducing malnutrition and stunting in particular, with a combination of nutrition-specific and nutrition-sensitive interventions yielding better outcome. In spite of recognizing nutritional value of insects and the contribution of cricket to improved gut health, there is limited evidence on the benefit of cricket based complementary food in reducing stunting amongst infants and young children. This study aims to determine the effect of integrating two nutrition interventions (cricket enriched porridge with nutrition education) on the infant and young child growth (stunting status) and gut health in rural Kenya; Alego Usonga Sub-County in Siaya County. The study is based on a 2x2 factorial design among infants aged 6 months and target to assess the main and combined effect of the two interventions (nutrition education and cricket enriched porridge) on the infant and young child's stunting and gut health. The study has four arms namely: Control arm (CA) where the study participants receive the standard care comprising of the supercereal Corn Soy Blend Plus (CSB+) in amounts adjusted for age, Enriched nutrition arm (ENA) where they receive the improved complementary food enriched with cricket and optimized for all the benefits of the cricket in amounts adjusted for age, Nutrition education arm (NEdA) where they receive nutrition education and a Combined Nutrition Education and enriched nutrition (CEdNA). The required sample size (based on the following parameters: Number of groups: = 4, effect size = 0.2, significance level = 0.05, power of test = 80%) is 70 study participants per study arm yielding a total of 280.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6 months at the time of enrolment,
2. Hemoglobin (Hb) of ≥7 g/dl (not severely anemic) and
3. Height for Age (HAZ) ≥-3 Z scores (not severely stunted).

Exclusion Criteria:

1. Those obviously ill and need medical attention who are referred for care as per ministry of health protocol
2. Children strictly fed on formula feed with no breast feeding
3. Infants whose caregivers do not consent or don't commit to adhere to the feeding regimen prescribed

Ages: 6 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 284 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-01-16 (Actual); Study Completion 2024-01-16 (Actual)

PRIMARY OUTCOMES:
Stunting (Height/Length for age Z scores) | 8 months
  Children who are too short for their age according to WHO 2005 growth standards. Length/Height in cm and age in months will be converted to Z scores using WHO Anthro and the values used to categorize growth as per the WHO 2005 standards

SECONDARY OUTCOMES:
Gut health | Baseline
  the integrity of the gut measured from stool illustrated by the gut microbiota(microbiome),Myeloperoxidase enzyme levels(MPO) as indicator of tissue inflammation plus butyrate concentration, alpha-1-anti trypsin (ATT) and Neopterin (NEO) & and 13C stable isotope breath test measured by the time it takes to recover 50% of the stable isotope and also the amount of carbon dioxide produced in the first 90 minutes after the dose with the 13Carbon stable isotope
Dietary intake | Baseline for breast milk intake, monthly for 8 months for the rest of the dietary intake information
  Total dietary intake including breast milk intake measured by deuterium oxide technique

CONTACTS AND LOCATIONS:
Overall Officials: Silvenus O. Konyole, PhD, Principal Investigator — Masinde Muliro University of Science and Technology
Locations (1):
- Rwambwa Sub County Hospital, Siaya, Western, Kenya

REFERENCES:
- [Derived] Okeyo NO, Wille CE, Kiiru SM, Sigot AJ, Ng'ang'a J, Kinyuru J, Roos N, Konyole SO. Effect of Edible Cricket Enriched Complementary Porridge and Nutrition Education on Linear Growth of Children 6-14 Months in Siaya County, Kenya: A Randomized 2 x 2 Factorial Trial. Matern Child Nutr. 2026 Mar;22(1):e70156. doi: 10.1111/mcn.70156. PMID 41503750